CLINICAL TRIAL: NCT06999434
Title: Exploring the Utility of [18F]3F4AP for Demyelination Imaging
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Georges El Fakhri, Professor of Radiology and Biomedical Imaging and of Biomedical Informatics & Data Science, Yale University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2000039282; 7P41EB022544-08 (NIH); 7R01EB033582-03 (NIH); 7R01AG076153-03 (NIH); 1R01AG085561-01 (NIH)
Record Dates: First submitted 2025-05-15; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Demyelinating Disorders; MCI; Alzheimer's Disease (AD); MS (Multiple Sclerosis); SCI - Spinal Cord Injury; Spinal Radiculopathy
Keywords: 3F4AP; Demyelinating Disorders; MS; SCI; AD
MeSH Terms: conditions — Demyelinating Diseases; Alzheimer Disease; Multiple Sclerosis; Spinal Cord Injuries | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Healthy Control (Active Comparator): n = 30 - up to three PET scanning sessions.
  Interventions: Drug: [ 18F]3F4AP; Drug: [18F]MK6240; Drug: [11C]PIB
- Alzheimer's Disease (AD) (Experimental): n = 15 - up to three PET scanning sessions.
  Interventions: Drug: [ 18F]3F4AP; Drug: [18F]MK6240; Drug: [11C]PIB
- Mild Cognitive Impairment (MCI) (Experimental): n = 15 - up to three PET scanning sessions.
  Interventions: Drug: [ 18F]3F4AP; Drug: [18F]MK6240; Drug: [11C]PIB
- Multiple Sclerosis (MS) (Experimental): n = 15 - up to three PET scanning sessions.
  Interventions: Drug: [ 18F]3F4AP; Drug: [18F]MK6240; Drug: [11C]PIB
- Spinal Cord Injury (SCI) (Experimental): n = 15 - up to three PET scanning sessions.
  Interventions: Drug: [ 18F]3F4AP; Drug: [18F]MK6240; Drug: [11C]PIB
- Spinal radiculopathy (SR) (Experimental): n = 15 - up to three PET scanning sessions.
  Interventions: Drug: [ 18F]3F4AP; Drug: [18F]MK6240; Drug: [11C]PIB

INTERVENTIONS:
Drug: [ 18F]3F4AP — PET Scan #3
Drug: [18F]MK6240 — PET Scan #2
Drug: [11C]PIB — PET Scan #1

SUMMARY:
The overall objective is to obtain an assessment of the pharmacokinetics of [18F]3F4AP in healthy volunteers and subjects with demyelinating diseases such as mild cognitive impairment (MCI), Alzheimer's Disease (AD), Multiple Sclerosis (MS), Spinal Cord Injury (SCI) and Spinal radiculopathy (SR).

ELIGIBILITY:
Inclusion:

1. Male and Female subjects must be ≥18 and <90 years of age;
2. Able to understand and provide informed consent prior to study procedures
3. Must be in good health

Exclusion:

1. Less than 18 years of age;
2. Pregnant or breastfeeding;
3. Any significant systemic illness or unstable medical condition;
4. Pre-existing medical conditions or claustrophobic reactions;
5. Research-related radiation exposure exceeds current PET Center guidelines (i.e. 50 mSv in the prior 12 months);
6. History of a bleeding disorder or are currently taking anticoagulants.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2030-05-05 (Estimated); Study Completion 2030-05-05 (Estimated)

PRIMARY OUTCOMES:
Tracers volume of distribution (VT) | 5 years
  PET images measured with [ 18F]3F4AP will quantify demyelination, those obtained with [18F]MK6240 will quantify tau burden and those obtained with [11C]PiB will reflect amyloid burden.
  PET images acquired with [18F]3F4AP, [18F]MK6240 and [11C]PiB, will measure the tracers volume of distribution (VT).
Distribution volume ratio (DVR) | 5 years
  PET images acquired with [18F]3F4AP, [18F]MK6240 and [11C]PiB, will measure the tracers distribution volume ratio (DVR).
Binding potential (BPND) | 5 years
  PET images acquired with [18F]3F4AP, [18F]MK6240 and [11C]PiB, will measure the tracers binding potential (BPND).
Demyelination | 5 years
  [18F]3F4AP will be used to measure demyelination. On the MR images, after co-registration and alignment, signal from pre- and post-contrast T1-weighted images, T2-weighted image, ratio between T1- and T2-weighted images (T1/T2) will be calculated to assess demyelination and white matter lesion (WML) on MR sequences.
Tau burden | 5 years
  [18F]MK6240 will be used to measure Tau burden.
Amyloid burden | 5 years
  [11C]PiB will reflect amyloid burden.
Tracer rate constant | 5 years
  The tracer rate constant for transfer from arterial plasma to tissue K1 and relative delivery R1 will also be estimated using tracer kineticmodeling technique, to provide measures of cerebral perfusion or CBF.
Associations between imaging modalities and biomarkers. | 5 years
  The Pearson correlation coefficient r will be used to assess the strength of the linear correlations between outcome measures. A P value of 0.05 or less will be considered statistically significant.

SECONDARY OUTCOMES:
Measure of brain atrophy | 5 years
  T1 images segmented and parcellated using FreeSurfer will be used to calculate cortical volumes, including the total cortical volume but also the hippocampal volume and will serve as proxies for neocortical and allocortical atrophy.
Measure of cerebrovascular burden | 5 years
  volume of White matter hyperintensities (WMH) on T1 images or T2 images
Measure of White matter lesions (WML) | 5 years
  The total WML load score will be calculated as the sum of the frequency of lesions multiplied by their volume.
MR/MRSI images | 5 years
  Evaluated to determine the effect of pulse sequence parameters and/or hardware configuration on image quality. The images acquired with different pulse sequence parameters or MR hardware configurations will be compared. Comparison of the MR images entails comparing the result of specific image quality measures such as signal-to-noise ratio (SNR) and contrast-to-noise ratio (CNR) as well as the level of image artifacts

CONTACTS AND LOCATIONS:
Overall Officials: Georges El Fakhri, PhD, DABR, Principal Investigator — Yale University
Locations (1):
- Yale University PET Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No